CLINICAL TRIAL: NCT05710913
Title: Development of Machine Learning Models for the Prediction of BMI and Complications After Bariatric Surgery (CABS-Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Med Anas Taha (Other)
Collaborators: University of Basel (Other); GZO Hospital, Zürich, Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Dr. Med Anas Taha, Research Fellow, University of Basel
Organization: University of Basel (Other)
Other Study IDs: CABS
Record Dates: First submitted 2023-01-15; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Body Weight; Post-Op Complication; Anastomosis, Leaking; Hiatal Hernia; GERD; Internal Hernia; Mesenteric Hernia; Intussusception; Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive
Keywords: Bariatric Surgery; Machine learning; Clinical prediction modelling; Artificial intelligence
MeSH Terms: conditions — Body Weight; Postoperative Complications; Hernia, Hiatal; Gastroesophageal Reflux; Internal Hernia; Intussusception; Diabetes Mellitus, Type 2; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Study aims to develop machine learning models with the ability to predict patients' BMI and complications after Bariatric Surgery (CABS-Score).

This Study also aims to develop machine learning models with the ability to predict diabetic (DM II)patients' remission rate after Bariatric Surgery.

The service mentioned above will be publicly available as a web-based application

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bariatric surgery
* Patients >18 years

Exclusion Criteria:

* Patients <18 years
* Patients who cannot be followed up on for more than 6 month after surgery
* Patients who are unable to provide informed approval to participate according to each centre's rules will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complication after surgery | [Time Frame: From index surgery up to 3 months postoperatively]
Body mass Index (KG/m2) after surgery | [Time Frame: From index surgery up to 1 year postoperatively]
Diabetes mellitus type II remission rate postoperatively | [Time Frame: From index surgery up to 2 year postoperatively]

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel - Department of Biomedical Engineering, Basel, Switzerland